CLINICAL TRIAL: NCT02529904
Title: A Phase II, Open Label Study to Describe Immune & Transcriptional Responses to MF59 Adjuvanted Trivalent Influenza Vaccine (ATIV) in Healthy 13-24 Month Children and Adults 18-65 Years
Brief Title: ADITEC FLU 2 STUDY: Understanding the Genetics Basis for Immune Responses to Flu Vaccines in Children and Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Emory University (Other); VisMederi srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OVG 2015/02
Record Dates: First submitted 2015-08-07; First posted 2015-08-20 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2018-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluad vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MF59 - ATIV (Experimental): All child participants will receive 2 doses of the MF59-ATIV, with the doses separated by 28 days.
  Adult participants will receive one dose of MF59-ATIV.
  Interventions: Biological: MF59 - ATIV

INTERVENTIONS:
Biological: MF59 - ATIV — All child participants will receive 2 doses of the MF59-ATIV, with the doses separated by 28 days.
  Adult participants will receive one dose of MF59-ATIV.
  Other Names: Fluad vaccine

SUMMARY:
Influenza infection is related to significant morbidity and mortality in children. The trivalent inactive vaccine (TIV) has been documented to have poor immunogenicity in children and the live attenuated influenza vaccine (ATIV) although proven to have more efficacy is unable to be administered to children under 2 years old. The MF59 adjuvanted influenza vaccine as proven efficacy on reducing the rates of laboratory confirmed influenza, including in children.

The study aims to assess early gene transcriptional responses to priming and boosting with MF59-ATIV in children aged 13-24 months and adults aged 18 - 65 years, and to establish correlations with haemagglutination inhibition (HAI) titers. It will be an open label study with 90 healthy children allocated to 3 groups (groups 1, 2 and 3) and 30 healthy adults allocated to group 4.

DETAILED DESCRIPTION:
Influenza infection is related to significant morbidity and mortality in children. The commonly used trivalent inactive influenza vaccine (TIV) has been documented to have poor immunogenicity in children, particularly in those less than 2 years old. The live attenuated influenza vaccine (LAIV) has shown improved efficacy compared to TIV, however LAIV is unable to be administered to children under 2 years old and those with contraindications, hence an effective alternative is required.

The focus toward adjuvanted influenza vaccines for children, particularly the MF59 adjuvant, has shown promising results in relation to safety and efficacy. This study aims to further explore the MF59 adjuvanted influenza vaccine from a gene expression perspective using a systems biology approach and relate these findings to innate immune responses, immunogenicity and reactogenicity.

The MF-59 adjuvant was approved for human use in 1997 and was studied initially in the elderly and more recently in children as young as 6 months. MF59-ATIV (Fluad®, Gripguard® (France) and Chiromas® (Spain)) is approved in Europe for adults aged 65 years and over and has been administered to over 5000 children in clinical trials.

In a recent large study with over 4000 children aged 6 months to 72 months, MF59-ATIV significantly reduced rates of laboratory-confirmed influenza with an absolute efficacy of 86%, demonstrating this vaccine to be an effective option for vaccinating children less than 2 years old unable to have the live attenuated vaccine. Unpublished data from the ADITEC Flu pilot study conducted in 2012 (EudraCT Number: 2012-002443-26, Ethics Ref: OxREC C 12/SC/0407); a phase 2, randomised, open label study, also demonstrated increased immunogenicity and a relatively similar reactogenicity profile following ATIV immunisation compared to TIV.

This study will use a systems biology approach to identify early gene signatures that relate to common innate and adaptive immune pathways following priming and boosting with ATIV, and to correlate these results with HAI response in children and adults.The systems biology approach has been used previously in vaccine research to identify gene module expression, including studies focusing on description of gene expression following the yellow fever vaccine (YF-17D), LAIV and TIV in adults. The study aims to assess early gene transcriptional responses to priming and boosting with MF59-ATIV in children aged 13-24 months and adults aged 18 - 65 years, and to establish correlations with HAI titers. It will be an open label study with 90 healthy children allocated to 3 groups (groups 1, 2 and 3) and 30 healthy adults allocated to group 4. Each participant will have an initial visit where screening will be completed and informed consent taken. The participant will then be enrolled and allocated a study participant number at this time. This initial visit ('Screening visit') will occur within the 56 days prior to the first ATIV immunisation. Group allocation will occur at or after the screening visit. Each child will receive 2 doses of ATIV and adults will receive 1 dose. ATIV is not currently licensed for children, and looking to previous studies, ATIV has been given to children less than 36 months as two 0.25 ml injections 4 weeks apart, and we will follow that immunisation schedule in this study. The timing of blood samples to be taken during the study will differ for each group in order to minimise number of blood collections per child but still enable assessment of gene expression and immune response at multiple time points.

ELIGIBILITY:
Inclusion Criteria:

* Children:

  * The investigator believes that the parents/LAR(s) of the child can and will comply with requirements of the protocol (e.g. completion of electronic diary, understanding of study procedure, consent process, availability at visits) and have internet access for the duration of the study.
  * Written informed consent obtained from parent/LAR(s) of the subject
  * Age from 13 months up to 24 months (excluding 24 months + 0 days and older) at time of V1 (first immunisation visit)
  * Born to two caucasian parents
  * Participant is healthy as determined by medical history and clinical examination
  * Have received all the vaccines specified in the UK immunisation schedule

Adults:

* Written and informed consent obtained from participant
* Age from 18 years up to 65 years (excluding 65 yrs + 0 days and older)
* Caucasian
* Participant has internet access for the duration of the study
* Participant is healthy as determined by medical history and clinical examination

Exclusion Criteria:

* Children

  * Child in care
  * Use (or planned use) of any non-registered or investigational product in last 30 days
  * Previous influenza vaccination
  * Microbiologically proven influenza illness or treatment with antiviral medications
  * Confirmed or suspected egg allergy
  * Chronic serious medical conditions which may, in the opinion of the investigator, interfere with evaluation of study objectives e.g. chronic lung disease, chronic liver/renal disease, chronic renal failure chronic heart disease, congenital genetic syndromes (e.g. Trisomy 21).
  * Recommended for influenza vaccine in UK (eg. Children in clinical risk groups as specified by Public Health England)
  * Suspected or confirmed immunosuppressive or immunodeficiency conditions (including splenic dysfunction & HIV)
  * Autoimmune conditions e.g. Type 1/2 diabetes mellitus, thyroid disease, juvenile idiopathic arthritis etc
  * Bleeding disorders

Adults

* Use (or planned use) of any non-registered or investigational product in last 30 days
* Confirmed or suspected egg allergy
* Chronic serious medical conditions which may, in the opinion of the investigator, interfere with evaluation of study objectives e.g. chronic lung disease, chronic liver/renal disease, chronic renal failure chronic heart disease
* Prior receipt of the 2015/2016 influenza vaccine
* Recommended for influenza vaccine in UK (eg. in clinical risk groups as specified by Public Health England)
* Suspected or confirmed immunosuppressive or immunodeficiency conditions (including splenic dysfunction & HIV)
* Autoimmune conditions e.g. Type 1/2 diabetes mellitus, thyroid disease, juvenile idiopathic arthritis etc
* Bleeding disorders
* Pregnancy

Ages: 13 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Early gene transcriptional responses to immunization with MF59-ATIV | 113 days
  Differential gene expression following ATIV baseline and days 1 and 3 post initial immunisation (adults and children) and at the baseline and day 1 and 3 post boots immunization (children). Gene expression analysis will be done using pax gene tubes for isolation of RNA
Relationship between early gene transcriptional responses and haemagglutination inhibition (HAI) responses | 113 days
  HAI titers and HAI geometric mean titers (GMT) and the mean geometric increase in HAI at baseline and day 28 (adults and childrens) and day 56 (childrens only). HAI titers thresholds defined as: influenza A H1N1 >= 1:40; influenza A H3N2 >=1:110; influenza b >= 1:620.

SECONDARY OUTCOMES:
Relationship between innate immune and gene transcriptional responses to ATIV immunization | 113 days
  Analysis of the frequency and activation of granulocytes, monocytes and dendritic cells as measured I the peripheral whole blood at the following time points: baseline and days 1,3 and 28 days post initial immunisation (adults and children) and at a day 1 and 3 post-boost immunisation (children)
Immunogenicity of ATIV in terms of HAI responses to each of the 3 vaccine strains | 113 days
  Percentage of participants with HAI titers (for strains influenza A H1N1, influenza A H3N2 and influenza B) defined as thresholds (1:40, 1:110 and 1:620), the HAI geometric mean titers (GMT) and the mean geometric increase in the HAI titers from baseline to day 28 (adults and children) and 56 (children)
Relationship between reactogenecity of ATIV (with particular focus on early inflammatory responses and early innate immune responses and gene transcriptional patterns | 113 days
  Percentage of participants experiencing local injection site adverse events (erythema (absent to severe (>=5 cm)), tenderness (none (0) to severe (3)), swelling (absent to severe (>=5 cm)), and systemic adverse events (for children: reduce feeding, reduced activity, increase irritability vomiting and diarrhoea (scores from none(0) to severe (3)); Adults: headache, nausea/vomiting, malaise, myalgia, arthralgia (scores from none (0) to severe (3)) around the time of the initial immunization (children and adults) and boost immunization (children)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Oxford, United Kingdom

REFERENCES:
- See also: Memory-like innate response to booster vaccination with MF-59 adjuvanted influenza vaccine in children — https://www.nature.com/articles/s41541-023-00702-1